CLINICAL TRIAL: NCT05468242
Title: A Phase II Trial of Tislelizumab as Consolidation Therapy in Patients With Locally Advanced Non-Small Cell Lung Cancer Who Have Not Progressed Following Neoadjuvant Chemotherapy Plus Tislelizumab ± Bevacizumab and Definitive Concurrent Chemoradiation Therapy
Brief Title: Study of Tislelizumab for Locally Advanced Non-Small Cell Lung Cancer Following Neoadjuvant Chemotherapy Plus Tislelizumab ± Bevacizumab and Definitive Concurrent Chemoradiation Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1086
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Stage III Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Radiotherapy; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant Chemotherapy Plus Tislelizumab + Bevacizumab (Experimental): Patients in experimental group will receive Tislelizumab consolidation (200 mg/q3w) after the neoadjuvant chemotherapy plus Tislelizumab + Bevacizumab and concurrent chemoradiotherapy.
  Interventions: Drug: Neoadjuvant chemo-immunotherapy; Drug: Bevacizumab; Radiation: Radiotherapy; Drug: Tislelizumab
- Neoadjuvant Chemotherapy Plus Tislelizumab (Active Comparator): Patients in this group will receive Tislelizumab consolidation (200 mg/q3w) after the neoadjuvant chemotherapy plus Tislelizumab and concurrent chemoradiotherapy.
  Interventions: Drug: Neoadjuvant chemo-immunotherapy; Radiation: Radiotherapy; Drug: Tislelizumab

INTERVENTIONS:
Drug: Neoadjuvant chemo-immunotherapy — The neoadjuvant chemo-immunotherapy before radiotherapy comprised of chemotherapy plus Tislelizumab [200 mg, once every 3 weeks (Q3W)].
Drug: Bevacizumab — The Bevacizumab was administrated concurrently with neoadjuvant chemo-immunotherapy (7.5mg/kg) once every 3 weeks (Q3W).
  Arms: Neoadjuvant Chemotherapy Plus Tislelizumab + Bevacizumab
Radiation: Radiotherapy — Definitive radiotherapy to the thoracic lesions.
Drug: Tislelizumab — Tislelizumab consolidation (200 mg) is performed once every 3 weeks after the neoadjuvant therapy and concurrent chemo-radiotherapy, and will continue on a Q3W schedule for a maximum duration of 12 months.

SUMMARY:
The phase II Study is to explore the efficacy and safety of Tislelizumab as consolidation therapy in patients with locally advanced non-small cell lung cancer who have not progressed following neoadjuvant chemotherapy plus Tislelizumab ± Bevacizumab and definitive concurrent chemoradiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in neoadjuvant therapy, patients should fulfil the following criteria:

  * Provision of signed, written and dated informed consent prior to any study specific procedures;
  * Male or female aged 18~75 years old;
  * Patients must have histologically- or cytologically-documented NSCLC who present with locally advanced (Stage III) disease;
  * Without prior chemotherapy, radiotherapy, surgery, targeted therapy or immunotherapy;
  * A recent tumour biopsy (taken following completion of the most recent therapy) is an optional requirement, provided that a biopsy procedure is technically feasible and the procedure is not associated with unacceptable clinical risk;
  * Life expectancy ≥12 weeks;
  * World Health Organization (WHO) Performance Status of 0 or 1;
  * Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients within 14 days before the use of study drug (HCG has a minimum sensitivity of 25 IU/L or equivalent);
  * Women must be non-breastfeeding
  * Forced expiratory volume in 1 second (FEV1) ≥800ml
  * Absolute neutrophil count >1.5 x 109/L (1500 per mm3)
  * Platelets >100 x 109/L (100,000 per mm3)
  * Haemoglobin≥9.0 g/dL (5.59 mmol/L)
  * Serum creatinine clearance(CL) >50 mL/min by the Cockcroft-Gault formula (Cockcroft and -Gault 1976)
  * Serum bilirubin ≤1.5 x upper limit of normal (ULN). Aspartate Transaminase(AST) and Alanine Transaminase(ALT) ≤2.5 x ULN

Exclusion Criteria:

* Exclusion criteria for enrolment for neoadjuvant therapy Patients should not enter the study if any of the following exclusion criteria are fulfilled:

  * Concurrent enrolment in another clinical study, unless it is an observational(non-interventional) clinical study;
  * Mixed small cell and non-small cell lung cancer histology;
  * Current or prior use of immunosuppressive medication within 28 days before the first dose of Tislelizumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Systemic steroid administration required to manage toxicities arising from radiation therapy delivered as part of the chemoradiation therapy for NSCLC is allowed.
  * Prior exposure to any anti-programmed cell death protein(PD)-1 or anti-PD-L1 antibody;
  * Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) that would prevent administration of Tislelizumab;
  * Active or prior documented autoimmune disease within the past 2 years;
  * Active or prior documented inflammatory bowel disease (eg. Crohn's disease, ulcerative colitis);
  * History of primary immunodeficiency;
  * History of organ transplant that requires therapeutic immunosuppression;
  * The tumor has completely approached, encircled, or invaded the intravascular space of the great vessels (e.g., the pulmonary artery or the superior vena cava)
  * Bleeding tendency or coagulation disorder
  * Hypertensive crisis, hypertensive encephalopathy, symptomatic heart failure (New York class II or above), active cerebrovascular disease or cardiovascular disease occurred within 6 months
  * Uncontrolled hypertension (systolic > 150mmHg and/or diastolic > 100mmHg)
  * Major surgery within 28 days or minor surgery or needle biopsy within 48 hours
  * Urine protein 3-4+, or 24h urine protein quantitative >1g
  * Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Bazett's Correction;
  * Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent;
  * Known history of tuberculosis;
  * Receipt of live attenuated vaccination within 30 days prior to study entry or within30 days of receiving Tislelizumab;
  * History of another primary malignancy within 5 years prior to starting Tislelizumab, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ and the disease under study;
  * Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control;
  * Any condition that, in the opinion of the investigator, would interfere with evaluation of the Tislelizumab or interpretation of patient safety or study results.
* Exclusion criteria for concurrent chemoradiation following neoadjuvant therapy

Patients should not enter the concurrent chemoradiation phase if any of the following exclusion criteria are fulfilled:

* Patients who develop disease progression and the irradiation dose of normal tissue will exceed the limit as defined in Section 7.
* World Health Organization (WHO) Performance Status of 2-4;
* Inadequate organ and marrow function as defined below:
* Forced expiratory volume in 1 second (FEV1) <800ml
* Absolute neutrophil count <1.5 x 109/L (1500 per mm3)
* Platelets <100 x 109/L (100,000 per mm3)
* Haemoglobin<9.0 g/dL (5.59 mmol/L)
* Serum creatinine CL <50 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976)
* Serum bilirubin >1.5 x upper limit of normal (ULN).
* Aspartate Transaminase(AST) and Alanine Transaminase(ALT) >2.5 x ULN

  * Further exclusion criteria for Tislelizumab consolidation:

Patients should not enter the Tislelizumab consolidation if any of the following exclusion criteria are fulfilled:

* Patients who have progressed whilst definitive platinum based, concurrent chemoradiation therapy;
* Current or prior use of immunosuppressive medication within 28 days before the first dose of Tislelizumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Systemic steroid administration required to manage toxicities arising from radiation therapy delivered as part of the chemoradiation therapy for locally advanced NSCLC is allowed.
* Any unresolved toxicity CTCAE >Grade 2 from the prior chemoradiation therapy will be excluded from randomization;
* Patients with Grade ≥2 pneumonitis from prior chemoradiation therapy will be excluded from randomization; Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE>Grade 1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2-year
  From the start date of initial treatment to progression, death or last follow-up.

SECONDARY OUTCOMES:
Overall survival | 2-year
  From the start date of initial treatment to death or to last follow-up.
Adverse Event | 2-year
  Toxicities were evaluated using the CTCAE 5.0
Health-related Quality of Life | 2-year
  An individual's or perceived physical and mental health during and after treatment.
Objective response rate | 2-year
  Tumor response to neoadjuvant immuno-chemotherapy and radiotherapy based on RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bezjak A, Temin S, Franklin G, Giaccone G, Govindan R, Johnson ML, Rimner A, Schneider BJ, Strawn J, Azzoli CG. Definitive and Adjuvant Radiotherapy in Locally Advanced Non-Small-Cell Lung Cancer: American Society of Clinical Oncology Clinical Practice Guideline Endorsement of the American Society for Radiation Oncology Evidence-Based Clinical Practice Guideline. J Clin Oncol. 2015 Jun 20;33(18):2100-5. doi: 10.1200/JCO.2014.59.2360. Epub 2015 May 5. PMID 25944914
- [Result] Machtay M, Bae K, Movsas B, Paulus R, Gore EM, Komaki R, Albain K, Sause WT, Curran WJ. Higher biologically effective dose of radiotherapy is associated with improved outcomes for locally advanced non-small cell lung carcinoma treated with chemoradiation: an analysis of the Radiation Therapy Oncology Group. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):425-34. doi: 10.1016/j.ijrobp.2010.09.004. Epub 2010 Oct 25. PMID 20980108
- [Result] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Result] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Result] Provencio M, Nadal E, Insa A, Garcia-Campelo MR, Casal-Rubio J, Domine M, Majem M, Rodriguez-Abreu D, Martinez-Marti A, De Castro Carpeno J, Cobo M, Lopez Vivanco G, Del Barco E, Bernabe Caro R, Vinolas N, Barneto Aranda I, Viteri S, Pereira E, Royuela A, Casarrubios M, Salas Anton C, Parra ER, Wistuba I, Calvo V, Laza-Briviesca R, Romero A, Massuti B, Cruz-Bermudez A. Neoadjuvant chemotherapy and nivolumab in resectable non-small-cell lung cancer (NADIM): an open-label, multicentre, single-arm, phase 2 trial. Lancet Oncol. 2020 Nov;21(11):1413-1422. doi: 10.1016/S1470-2045(20)30453-8. Epub 2020 Sep 24. PMID 32979984
- [Result] Herbst RS, Giaccone G, de Marinis F, Reinmuth N, Vergnenegre A, Barrios CH, Morise M, Felip E, Andric Z, Geater S, Ozguroglu M, Zou W, Sandler A, Enquist I, Komatsubara K, Deng Y, Kuriki H, Wen X, McCleland M, Mocci S, Jassem J, Spigel DR. Atezolizumab for First-Line Treatment of PD-L1-Selected Patients with NSCLC. N Engl J Med. 2020 Oct 1;383(14):1328-1339. doi: 10.1056/NEJMoa1917346. PMID 32997907
- [Result] Zhang YQ, Hu PC, Wu RZ, Gu YS, Chen SG, Yu HJ, Wang XQ, Song J, Shi HC. The image quality, lesion detectability, and acquisition time of 18F-FDG total-body PET/CT in oncological patients. Eur J Nucl Med Mol Imaging. 2020 Oct;47(11):2507-2515. doi: 10.1007/s00259-020-04823-w. Epub 2020 May 18. PMID 32424483